CLINICAL TRIAL: NCT03265301
Title: Corrective Office Hysteroscopic Surgery Versus Conventional Hysteroscopy in Treatment of Intrauterine Abnormalities
Brief Title: Hysteroscopic Surgery in Treatment of Intrauterine Abnormalities
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The randomization could not be done
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSIU
Record Dates: First submitted 2017-08-27; First posted 2017-08-29 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Office hysteroscopy (Other)
  Interventions: Procedure: Hysteroscopy; Procedure: Office hysteroscopy
- Conventional hysteroscopy (Other)
  Interventions: Procedure: Hysteroscopy; Procedure: Conventional hysteroscopy

INTERVENTIONS:
Procedure: Hysteroscopy — Includes Video set up, mini-hysteroscope system, continuous inflow and outflow, rod lens or fiber optic lens Zero to 30 degree angle and mechanical instruments (Scissors,Graspers , Cup biopsy forceps and bipolar instruments)
Procedure: Office hysteroscopy — will be done in out patient clinic without anesthesia
  Arms: Office hysteroscopy
Procedure: Conventional hysteroscopy — will be done in operative room under general anesthesia
  Arms: Conventional hysteroscopy

SUMMARY:
With the ongoing developments in the field of hysteroscopy during the past 15 years, hysteroscopic surgery is becoming safer and less invasive for the patient. Improved technology has enabled surgeons to perform many operative procedures in an ambulatory setting without significant patient discomfort and with potentially significant cost savings.

Office operative hysteroscopy (see and treat hysteroscopy) reduces the distinction between a diagnostic and an operative procedure, shifting the focus in health care away from inpatient diagnosis and treatment. The development of smaller-diameter hysteroscopes with continuous-flow system features and working channels, through which operative instruments can be introduced, has made it possible to treat some uterine and cervical diseases without the traditional need for cervical dilation or general anesthesia.

Use of specially designed hysteroscopic 5F mechanical instruments (e.g., scissors, biopsy cup, graspers, and corkscrews) has long been the only way to perform operative procedures in an ambulatory setting. However, although grasping forceps and scissors are excellent for treating adhesions, cervical polyps, and endometrial polyps smaller than or the same size as the larger endometrial polyps, or thick lesions (e.g., submucous fibroids) were difficult to treat successfully using such miniature, fragile instruments and without cervical dilation.

An important technologic advance occurred in 1997 with the introduction of a versatile bipolar electrosurgery system dedicated to hysteroscopy, the Gynecare VersaPoint (Ethicon, Inc., Somerville, NJ, USA), which represents a key point in the history of office operative hysteroscopy. With the use of 5F bipolar electrodes, the number of pathologic conditions treated using office operative hysteroscopy has increased tremendously, reducing the use of the resectoscope and the operating room to a smaller number of cases.

More recently, a new generation of electrical generators, allowing the use of bipolar energy on miniaturized electrodes, has been presented (Autocon 400 II; Karl Storz Endoscopy, Tuttlingen, Germany). The main advantage of these instruments is that they are reusable, thereby reducing the costs of office operative as those described for the Versapoint system.

The feasibility of ambulatory uterine surgery is not just dependent on recent technological advances in instrumentation such as miniaturization of equipment, but also the favorable anatomical characteristics of the uterus itself. The sensitive innervations of the uterus originate in the myometrium and extend to the outer serosal surface, whereas the endometrium and any fibrotic tissue within the cavity are less sensitive. Thus, procedures can be carried out without the use of analgesia or anesthesia.

However, a careful operative technique is of paramount importance, in particular, avoiding inadvertent deep penetration of the superficial myometrium when resecting lesions such as polyps, maintaining the lowest possible distension pressures, and expediting procedures through efficient surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* infertile women
* women with recurrent pregnancy loss
* suspected intrauterine abnormalities

Exclusion Criteria:

* Normal endometrial cavity
* Endometrial pathologies like polypi or submucous myomata.
* Extensive intrauterine synechiae

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Number of uterine abnormalities which will be treated successfully by office and conventional hysteroscopy | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided